CLINICAL TRIAL: NCT03433820
Title: A Single-arm, Observational Study to Explore and Characterize Wound Healing After Skin Punch Biopsies in Healthy Volunteers
Brief Title: Wound Healing in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Human Drug Research, Netherlands (Other)
Collaborators: Maruho Co., Ltd. (Industry)
Responsible Party: Principal Investigator, prof dr J. Burggraaf, Research Director, Centre for Human Drug Research, Netherlands
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHDR1736
Record Dates: First submitted 2018-01-23; First posted 2018-02-15 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Wound Healing
MeSH Terms: interventions — Wound Healing

STUDY DESIGN:
Intervention Model Description: A single-arm, observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- randomized repeated biopsy (Experimental): The study will entail 1 cohort with a randomized repeated biopsy collection time. Three skin punch biopsies (3 mm) of the lower back will be taken from each volunteer on day 0. One biopsy sample taken on day 0 will serve as a baseline measurement for the repeated samples regarding the histology, immunohistochemistry, and RNA sequencing (RNA-seq) or real-time reverse transcription polymerase chain reaction (qRT-PCR) assessments.
  Repeated biopsies of the same location as on day 0 will be taken on day 7, 14 or 21 (biopsy lesion and day randomized), and day 28, 42 or 56 (biopsy lesion and day randomized) for all subjects. The observation biopsy (biopsy lesion randomized) will serve as primary biopsy and followed for all measurements.
  Interventions: Other: Observation of wound healing

INTERVENTIONS:
Other: Observation of wound healing — Observation of wound healing after skin biopsy

SUMMARY:
The skin plays a critical role in protection where it acts as a barrier from damage and pathogens between the external and internal environments. Wounds compromise its protective role by disrupting the function and the normal structure of the skin and the underlying soft tissue. As a response to injury wound healing occurs in order to rapidly restore the defect. This process involves activation of keratinocytes, fibroblasts, endothelial cells, macrophages, and platelets and consists of multiple phases including hemostasis, inflammation, migration and cellular proliferation, and maturation and remodeling. A simplified schematic of the course of wound healing is depicted in Figure 2. Hemostasis occurs immediately after dermal injury. The inflammation phase is characterized by cellular recruitment and increased vascular permeability. The epithelization phase is achieved by proliferation of basal cells and migration of epithelial cells. The last phase is known as the maturation and remodeling phase where collagen cross-linking and remodeling, wound contraction, and repigmentation takes place. Due to the broad involvement of various cell types, extracellular matrix and many reactive molecules each phase in wound healing produces characteristic changes within the tissue. A deficiency in any part of the process can lead to delayed wound healing, abnormal scar formation or chronic wounds.

To study wound healing in healthy volunteers a challenge model with skin punch biopsies has been described in literature previously. However, the characterization of this model was not performed comprehensively since advanced analysis of biopsies were omitted. Furthermore, analyses performed in previous studies only partially described wound healing processes either by insufficient time points for characterization or scarce simultaneous evaluations of multiple wound healing modalities.

The overall aim of this study is to develop a standardized model to temporarily and locally induce a skin trauma to investigate wound healing and monitor wound closure. This clinical model will enable future application as proof-of-pharmacology and proof-of concept studies as well as drug profiling in early drug development programs. More specifically, the objective of the trial is to explore and characterize the induction of well-defined skin trauma and natural wound healing process over the course of the different phases using a battery of dermatological assessments after skin punch biopsies in healthy volunteers. Furthermore, safety and tolerability will be assessed.

Characterization and monitoring of wound healing effects following skin punch biopsies will be performed by means of biophysical, biochemical, imaging, clinical parameters and subject reported outcomes.

DETAILED DESCRIPTION:
Background & Rationale The skin plays a critical role in protection where it acts as a barrier from damage and pathogens between the external and internal environments. Wounds compromise its protective role by disrupting the function and the normal structure of the skin and the underlying soft tissue. As a response to injury wound healing occurs in order to rapidly restore the defect. This process involves activation of, among others, keratinocytes, fibroblasts, endothelial cells, macrophages, and platelets and consists of multiple phases including hemostasis, inflammation, migration and cellular proliferation, and maturation and remodeling. A simplified schematic of the course of wound healing is depicted in Figure 2. Due to the broad involvement of various cell types, extracellular matrix and many reactive molecules each phase in wound healing produces characteristic changes within the tissue. A deficiency in any part of the process can lead to delayed wound healing, abnormal scar formation or chronic wounds.

To study wound healing in healthy volunteers a challenge model with skin punch biopsies has been described in literature previously. However, the characterization of this model was not performed comprehensively since advanced analysis of biopsies were omitted. Furthermore, analyses performed in previous studies only partially described wound healing processes either by insufficient time points for characterization or scarce simultaneous evaluations of multiple wound healing modalities. In addition, novel non-invasive imaging methodologies including thermography, 3D photography, multispectral imaging, enable more comprehensive profiling of the wound morphology.

The overall aim of this study is to develop a standardized model to temporarily and locally induce a skin trauma to investigate wound healing and monitor wound closure. This clinical model will enable future application as proof-of-pharmacology and proof-of concept studies as well as drug profiling in early drug development programs. More specifically, the objective of the trial is to explore and characterize the induction of well-defined skin trauma and natural wound healing process over the course of the different phases using a battery of dermatological assessments after skin punch biopsies in healthy volunteers. Furthermore, safety and tolerability will be assessed.

Characterization and monitoring of wound healing effects following skin punch biopsies will be performed by means of biophysical, biochemical, imaging, clinical parameters and subject reported outcomes.

Objective(s) Primary Objective

* To characterize and monitor wound healing after a standardized, induced skin trauma Secondary Objectives
* To evaluate safety and tolerability of biopsy-induced skin trauma Design This is an observational, single center, single arm study. Treatments Biopsy sites will be treated by secondary healing intention with a non-stick gauze dressing followed by no treatment after 48h.

Investigational drug Not applicable Comparative drug No comparative drug will be used in this study. Study periods The total duration of the study will be approximately 14 weeks: 4 weeks for screening and 10 weeks of observation. Subjects will visit CHDR 14 times.

Subjects / Groups A total of 18 healthy volunteers are planned to be enrolled. The study will entail 1 cohort with a randomized repeated biopsy collection time. Three skin punch biopsies (3 mm) of the lower back will be taken from each volunteer on day 0, with a distance of approximately 3-5 cm in between. All biopsy lesions will be treated with a gauze dressing (Jelonet®, paraffine gauze + Tegaderm®) for 48h after which the gauze is removed. Hereafter, the biopsy lesions will remain untreated. One biopsy sample taken on day 0 will serve as a baseline measurement for the repeated samples regarding the histology, immunohistochemistry, and RNA sequencing (RNA-seq) or real-time reverse transcription polymerase chain reaction (qRT-PCR) assessments.

Repeated biopsies of the same location as on day 0 will be taken on day 7, 14 or 21 (biopsy lesion and day randomized), and day 28, 42 or 56 (biopsy lesion and day randomized) for all subjects. The observation biopsy (biopsy lesion randomized) will serve as primary biopsy and followed for all measurements. All repeated biopsy lesions will also be treated with a gauze dressing (Jelonet®, paraffine gauze + Tegaderm®) for 48h after which the gauze is removed and observation commences.

Cohort: 1 Observation period (day 2 - day 70): 3 biopsies taken on day 0

* 1 repeated biopsy taken on day 7, 14 or 21 (randomized)
* 1 repeated biopsy taken on day 28, 42 or 56 (randomized)
* 1 target (primary) biopsy for observation without re-excision Number of subjects: 18

Inclusion criteria

Eligible subjects must meet all of the following inclusion criteria at screening:

1. Healthy subjects, 18 to 30 years of age (inclusive). The health status is verified by absence of evidence of any clinical significant active or uncontrolled chronic disease following a detailed medical history, a complete physical examination including vital signs, blood sampling of hematology, chemistry, and virology, urinalysis, urine drug and cotinine testing, and alcohol breath testing. In the case of uncertain or questionable results, tests performed during screening may be repeated before randomization to confirm eligibility or judged to be clinically irrelevant for healthy subjects.
2. Body mass index (BMI) between 18 and 30 kg/m2, inclusive
3. Fitzpatrick Skin type I-II (Caucasian type).
4. Eligible lower back to perform biopsies (no excessive hair growth, no local skin disorder)
5. Willing to give written informed consent and willing and able to comply with the study protocol.

Exclusion criteria

Eligible subjects must meet none of the following exclusion criteria at screening:

1. History of pathological scar formation (keloid, hypertrophic scars)
2. Any form of body modification of the lower back hindering biopsy collection of unaltered skin (e.g. tattoos, piercings, implants)
3. Any disease associated with immune system impairment, including auto-immune diseases, HIV and transplantation patients.
4. Requirement of immunosuppressive or immunomodulatory medication, including glucocorticoids, non-steroid anti-inflammatory drugs (NSAIDs), and chemotherapeutic drugs within 30 days prior to enrollment or planned to use during the course of the study.
5. Have any current and/or recurrent pathologically, clinical significant relevant skin condition.
6. Use of topical medication (prescription or over-the-counter (OTC)) within 30 days of the start of the study.in local treatment area.
7. Pregnant, a positive pregnancy test, intending to become pregnant, or breastfeeding.
8. Current smoker and/or regular user of other nicotine-containing products (e.g., patches).
9. Average consumption of more than 14 units of alcohol per week
10. Tanning due to sunbathing, excessive sun exposure or a tanning booth within 3 weeks of enrollment or planned to do so during the course of the study
11. Participation in an investigational drug or device study within 3 months prior to screening or more than 4 times a year.
12. Loss or donation of blood over 500 mL within three months prior to screening.
13. Any (medical) condition that would, in the opinion of the investigator, potentially compromise the safety or compliance of the subject or may preclude the subjects' successful completion of the clinical trial.

Concomitant medications No prescription medication or OTC medications (excluding multivitamins) will be permitted within 21 days prior to the start of the study, or less than 5 half-lives (whichever is longer), and during the course of the study. Exceptions are paracetamol (up to 4 g/day) in case of local pain. Use of pain medication will be determined by the investigator individually. Other exceptions will only be made if the rationale is discussed and clearly documented.

Endpoints

* Biopsy biomarkers:

  * Histology with hematoxylin and eosin (HE) staining
  * Immunohistochemistry with wound healing related biomarkers (e.g. CD31, collagen I, collagen III, aSMA, fibronectin)
  * RNA-seq or qRT-PCR for wound healing related biomarkers (e.g. VEGFα, TGFβ1, TGFβ2, TGFβ3, PDGF, CTGF, TNF, IL-1B, IL-4, GM-CSF, IL-6, IL-10, MMP1, MMP3, OSM, LOX)
* Local skin biomarkers for wound healing related biomarkers (e.g. VEGF-A, TNFα, IL-8, TLSP, MMP-3, IL-4) by transdermal analysis patch (TAP)
* Clinical imaging (e.g. 2D and 3D photography, thermography, laser speckle contrast imaging (LSCI), trans epidermal water loss (TEWL), colorimetry)
* Clinical evaluation (erythema grading scale, Red-Yellow-Black (RYB) wound assessment scale, the Patient and Observer Scar Assessment Scale (POSAS))
* Skin microbiome (healthy and biopsy lesions) Tolerability / safety endpoints
* Adverse events (AEs)
* Local tolerance (erythema grading scale, RYB wound assessment scale, POSAS, NRS pruritus and pain) All of above mentioned pharmacodynamic and safety measurements will be performed multiple times during the study according to the Visit and assessment schedule.

Sample Size Justification A total cohort size of 18 healthy volunteers will be investigated. This is justified since the primary objective is to explore and monitor the wound healing model. No formal power calculation was performed given the exploratory character of the study.

Statistical methodology Data listings and averages will be presented for pharmacodynamics and safety measures.

Given the exploratory character of the study, pharmacodynamic endpoints will be primarily analyzed using descriptive statistics. All pharmacodynamic endpoints will be summarized (mean and standard deviation of the mean, median, minimum and maximum values) by time, and will also be presented graphically as mean over time, with standard deviation as error bars. Both Nominal results, and log-transformed results and change from baseline results will be utilized in all data summaries. All categorical pharmacodynamic endpoints will be summarized by frequencies.

ELIGIBILITY:
Inclusion criteria

Eligible subjects must meet all of the following inclusion criteria at screening:

1. Healthy subjects, 18 to 30 years of age (inclusive). The health status is verified by absence of evidence of any clinical significant active or uncontrolled chronic disease following a detailed medical history, a complete physical examination including vital signs, blood sampling of hematology, chemistry, and virology, urinalysis, urine drug and cotinine testing, and alcohol breath testing. In the case of uncertain or questionable results, tests performed during screening may be repeated before randomization to confirm eligibility or judged to be clinically irrelevant for healthy subjects.
2. Body mass index (BMI) between 18 and 30 kg/m2, inclusive
3. Fitzpatrick Skin type I-II (Caucasian type).
4. Eligible lower back to perform biopsies (no excessive hair growth, no local skin disorder)
5. Willing to give written informed consent and willing and able to comply with the study protocol.

Exclusion criteria

Eligible subjects must meet none of the following exclusion criteria at screening:

1. History of pathological scar formation (keloid, hypertrophic scars)
2. Any form of body modification of the lower back hindering biopsy collection of unaltered skin (e.g. tattoos, piercings, implants)
3. Any disease associated with immune system impairment, including auto-immune diseases, HIV and transplantation patients.
4. Requirement of immunosuppressive or immunomodulatory medication, including glucocorticoids, non-steroid anti-inflammatory drugs (NSAIDs), and chemotherapeutic drugs within 30 days prior to enrollment or planned to use during the course of the study.
5. Have any current and/or recurrent pathologically, clinical significant relevant skin condition.
6. Use of topical medication (prescription or over-the-counter (OTC)) within 30 days of the start of the study.in local treatment area.
7. Pregnant, a positive pregnancy test, intending to become pregnant, or breastfeeding.
8. Current smoker and/or regular user of other nicotine-containing products (e.g., patches).
9. Average consumption of more than 14 units of alcohol per week
10. Tanning due to sunbathing, excessive sun exposure or a tanning booth within 3 weeks of enrollment or planned to do so during the course of the study
11. Participation in an investigational drug or device study within 3 months prior to screening or more than 4 times a year.
12. Loss or donation of blood over 500 mL within three months prior to screening.
13. Any (medical) condition that would, in the opinion of the investigator, potentially compromise the safety or compliance of the subject or may preclude the subjects' successful completion of the clinical trial.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 18 to 30 years of age (inclusive)
Enrollment: 18 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Biopsy biomarkers | 3 months after end of study
  Histology with hematoxylin and eosin (HE) staining
Local skin biomarkers | 3 months after end of study
  Local skin biomarkers for wound healing related biomarkers (e.g. VEGF-A, TNFα, IL-8, TLSP, MMP-3, IL-4) by transdermal analysis patch (TAP)
Clinical imaging | 3 months after end of study
  2D photography
Clinical evaluation | 3 months after end of study
  Erythema grading scale. Wounds are scored on the basis of redness of the wound (from better to worse: absence, mild, moderate, or severe).
Skin microbiome | 3 months after end of study
  Skin microbiome (healthy and biopsy lesions). Collection of skin culture samples is a non-invasive procedure where a sterile polyester flock tip per site is passed along the surface of the 3 different areas. The target areas are i) regions surrounding one of the biopsy lesions on the lower back, ii) a control site of healthy, unaffected skin in proximity of a biopsy lesion and iii) a control area on the lower back with a minimum distance of 10cm from a biopsy site. The skin swab will be placed in a 2 ml lysis tube containing DNA/RNA shield to stabilize and preserve the DNA. The DNA extraction will be performed using adapted DNA extraction method based on the Zymo Research fecal DNA extraction methodology. After DNA extraction, the variable regions 3 and 4 of the 16S rRNA gene are amplified giving an amplicon of around 450 base pairs. This amplicon is analyzed by capillary systems using standard protocols.
Biopsy biomarkers | 3 months after end of study
  Immunohistochemistry with wound healing related biomarkers (e.g. CD31, collagen I, collagen III, aSMA, fibronectin)
Biopsy biomarkers | 3 months after end of study
  RNA-seq or qRT-PCR for wound healing related biomarkers (e.g. VEGFα, TGFβ1, TGFβ2, TGFβ3, PDGF, CTGF, TNF, IL-1B, IL-4, GM-CSF, IL-6, IL-10, MMP1, MMP3, OSM, LOX)
Clinical imaging | 3 months after end of study
  3D photography
Clinical imaging | 3 months after end of study
  Thermography
Clinical imaging | 3 months after end of study
  Laser speckle contrast imaging (LSCI)
Clinical imaging | 3 months after end of study
  Trans epidermal water loss (TEWL)
Clinical imaging | 3 months after end of study
  Colorimetry
Clinical evaluation | 3 months after end of study
  Red-Yellow-Black (RYB) wound assessment scale. Wounds are scored based on the color of the wound bed (from healthy to least healthy: red, yellow, or black). The least healthy color is chosen in multi-color wounds. Furthermore, a humidity subscale (dry, humid, or wet) is added to further classify the health status of the wounds.
Clinical evaluation | 3 months after end of study
  POSAS. The observer scale of the POSAS consists of six items (vascularity, pigmentation, thickness, relief, pliability and surface area). All items are scored on a scale ranging from 1 ('like normal skin') to 10 ('worst scar imaginable'). The sum of the six items results in a total score of the POSAS observer scale. Categories boxes are added for each item:
  * Vascularity category: pale, pink, red, purple, mix
  * Pigmentation category: hypo, hyper, mix
  * Thickness category: thicker, thinner
  * Relief category: more, less, mix
  * Surface area category: expansion, contraction, mix Furthermore, an overall opinion is scored on a scale ranging from 1 to 10. All parameters are preferably compared to normal skin on a comparable anatomic location.

SECONDARY OUTCOMES:
Adverse events (AEs) | 3 months after end of study
  Adverse events
Local tolerance | 3 months after end of study
  Erythema grading scale. Wounds are scored on the basis of redness of the wound (from better to worse: absence, mild, moderate, or severe).
Local tolerance | 3 months after end of study
  Red-Yellow-Black (RYB) wound assessment scale. Wounds are scored based on the color of the wound bed (from healthy to least healthy: red, yellow, or black). The least healthy color is chosen in multi-color wounds. Furthermore, a humidity subscale (dry, humid, or wet) is added to further classify the health status of the wounds.
Local tolerance | 3 months after end of study
  POSAS. The observer scale of the POSAS consists of six items (vascularity, pigmentation, thickness, relief, pliability and surface area). All items are scored on a scale ranging from 1 ('like normal skin') to 10 ('worst scar imaginable'). The sum of the six items results in a total score of the POSAS observer scale. Categories boxes are added for each item:
  * Vascularity category: pale, pink, red, purple, mix
  * Pigmentation category: hypo, hyper, mix
  * Thickness category: thicker, thinner
  * Relief category: more, less, mix
  * Surface area category: expansion, contraction, mix Furthermore, an overall opinion is scored on a scale ranging from 1 to 10. All parameters are preferably compared to normal skin on a comparable anatomic location.
Local tolerance | 3 months after end of study
  NRS pruritus and pain. The pruritus and pain NRS are single-question assessment tools that are used to assess the subject's worst itch and pain in the previous time interval. Subjects will be asked the following question; "on a scale of 0 - 100, with 0 being no itch, and 100 being the worst itch imaginable, how would you rate your average degree of itch of all biopsy sites combined experienced during the previous time interval?" and "on a scale of 0 - 100, with 0 being no pain, and 100 being the worst pain imaginable, how would you rate your average degree of pain of all biopsy sites combined experienced during the previous time interval?"

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rissmann, PhD, Principal Investigator — CHDR
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands

REFERENCES:
- [Background] Dreifke MB, Jayasuriya AA, Jayasuriya AC. Current wound healing procedures and potential care. Mater Sci Eng C Mater Biol Appl. 2015 Mar;48:651-62. doi: 10.1016/j.msec.2014.12.068. Epub 2014 Dec 19. PMID 25579968
- [Background] Greaves NS, Benatar B, Whiteside S, Alonso-Rasgado T, Baguneid M, Bayat A. Optical coherence tomography: a reliable alternative to invasive histological assessment of acute wound healing in human skin? Br J Dermatol. 2014 Apr;170(4):840-50. doi: 10.1111/bjd.12786. PMID 24329481
- [Background] Greaves NS, Iqbal SA, Hodgkinson T, Morris J, Benatar B, Alonso-Rasgado T, Baguneid M, Bayat A. Skin substitute-assisted repair shows reduced dermal fibrosis in acute human wounds validated simultaneously by histology and optical coherence tomography. Wound Repair Regen. 2015 Jul-Aug;23(4):483-94. doi: 10.1111/wrr.12308. Epub 2015 Jul 31. PMID 26053202
- [Background] Illigens BM, Gibbons CH. A human model of small fiber neuropathy to study wound healing. PLoS One. 2013;8(1):e54760. doi: 10.1371/journal.pone.0054760. Epub 2013 Jan 31. PMID 23382960
- [Background] Ud-Din S, Greaves NS, Sebastian A, Baguneid M, Bayat A. Noninvasive device readouts validated by immunohistochemical analysis enable objective quantitative assessment of acute wound healing in human skin. Wound Repair Regen. 2015 Nov-Dec;23(6):901-14. doi: 10.1111/wrr.12344. Epub 2015 Nov 4. PMID 26174693
- [Background] Ud-Din S, Perry D, Giddings P, Colthurst J, Zaman K, Cotton S, Whiteside S, Morris J, Bayat A. Electrical stimulation increases blood flow and haemoglobin levels in acute cutaneous wounds without affecting wound closure time: evidenced by non-invasive assessment of temporal biopsy wounds in human volunteers. Exp Dermatol. 2012 Oct;21(10):758-64. doi: 10.1111/exd.12005. PMID 23078397
- See also: Basic principles of wound healing — http://www.uptodate.com/contents/basic-principles-of-wound-healing

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/20/NCT03433820/Prot_SAP_000.pdf